CLINICAL TRIAL: NCT04471883
Title: Latin American Registry of Percutaneous Interventions in Coronary Bifurcations
Brief Title: LATAM Bif Registry
Status: Not yet recruiting | Type: Observational
Sponsor: LATAM Bifurcation Club (Network)
Responsible Party: Sponsor
Other Study IDs: 00543186
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Coronary Bifurcation Lesion
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous coronary interventions — Percutaneous coronary interventions in coronary bifurcation lesions

SUMMARY:
The LATAM Bif Registy is an international and prospective registry of percutaneous coronary interventions (PCI) in coronary bifurcation lesions. The main goal of the study is to investigate the current state and long-term outcomes of PCI in this complex subset of coronary lesions in Latin America.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Any type of bifurcation lesion
* Side-branch reference diameter >= 2 mm

Exclusion Criteria:

* Protected left main disease in patients with previous CABG
* Patients who refuse to be included in the registry

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients ≥18 years of age, who have at least one significant lesion in a coronary bifurcation on diagnostic cinecoronary angiography and who are candidates to treatment with PCI, regardless of the dedicated-technique used. Those patients who present lesions involving vessels <2 mm by visual estimation and those who refuse to be included in the registry will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Cardiac Death | 5 years
Myocardial Infarction | 5 years
Target Lesion Revascularization | 5 years
Stent thrombosis | 5 years
Major bleeding | 5 years

IPD SHARING:
Plan to Share IPD: No
No IPD planned